CLINICAL TRIAL: NCT06103578
Title: Evaluation of Gingival Crevicular Fluid and Saliva SOST and TWEAK, Gingival Crevicular Fluid RANKL and OPG Levels in Smokers and Non-smokers With Periodontitis
Brief Title: Evaluation of SOST, TWEAK, RANKL, OPG Levels in Smokers and Non-Smokers With Periodontitis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ece Güner, Assistant researcher, Gazi University
Other Study IDs: 6362
Record Dates: First submitted 2023-09-13; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis; Smoking
Keywords: periodontitis; smoking; RANKL; OPG; TWEAK; SOST
MeSH Terms: conditions — Periodontitis; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-smoker periodontitis
  Interventions: Diagnostic Test: GCF and saliva analysis
- Smoker periodontitis
  Interventions: Diagnostic Test: GCF and saliva analysis
- Control
  Interventions: Diagnostic Test: GCF and saliva analysis

INTERVENTIONS:
Diagnostic Test: GCF and saliva analysis — ELISA

SUMMARY:
Periodontitis is a chronic inflammatory disease with multifactorial etiology. Although periodontal disease is initiated by pathogens within the biofilm layer, disease development and tissue destruction occur as a result of the interaction of periodontal pathogens and the host immune response. It has been determined in the literature that smoking has a significant negative effect on periodontal tissues and increases the risk of periodontitis by 2-5 times. It has been shown that there is a relationship between smoking and the incidence and progression of periodontitis. However, the mechanisms by which this occurs have not been explained. In this study, the effect of smoking on the levels of sclerostin (SOST), tumor necrosis factor-like weak inducer of apoptosis (TWEAK), receptor activator of nuclear factor-kB ligand (RANKL), and osteoprotegerin (OPG), which are effective in bone metabolism, in gingival crevicular fluid (GCF) and saliva will be evaluated. Participants in the study were in accordance with the 2017 World Workshop on Classification of Periodontal and Peri-implant Diseases and Conditions criteria as a result of clinical evaluations systemically healthy, non-smokers diagnosed with stage 2, 3 and/or 4 periodontitis (Group 1) (n=26); systemically healthy, diagnosed with stage 2, 3 and/or 4 periodontitis and smokers (Group 2) (n=26); systemically and periodontally healthy, non-smokers (Group 3-Control Group) (n=26). Clinical periodontal indixes will be obtained from participants meeting the inclusion criteria; GCF and saliva samples will be collected. The samples will be examined by ELISA test at Gazi University Faculty of Medicine, Department of Immunology.

ELIGIBILITY:
Inclusion Criteria:

* Study participants have no history of periodontal therapy or drug therapy for at least 6 months.

Exclusion Criteria:

* Pregnancy, lactation, during orthodontic treatment and systemic conditions related to bone metabolism, diabetes were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Periodontitis: Stage 2,3,4 and grade A,B,C periodontitis non-smoker patient included.
  Smoking-periodontitis: Stage 2,3,4 and grade A,B,C periodontitis patients which smoking 10 or more daily for at least 10 years included.
  Control: Periodontally healthy, non-smoker subjects included.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Plaque index (Silness & Löe ) | Clinical periodontal indices were recorded at the participants' first visit.
  This index ascertains the thickness of plaque along the gingival margin. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. The scores from the four areas of the tooth are added and divided by four for each tooth score. When creating the whole mouth score, the arithmatic average of all tooth scores was taken.
Gingival index (Löe & Silness) | Clinical periodontal indices were recorded at the participants' first visit.
  Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. The scores from the four areas of the tooth are added and divided by four for each tooth score. When creating the whole mouth score, the arithmatic average of all tooth scores was taken.
Probing depth | Clinical periodontal indices were recorded at the participants' first visit.
  Probing depth is the distance from the gingival margin to the apical portion of the gingival sulcus. The scores from the four areas of the tooth are added and divided by four for each tooth score. It is recorded as mm. When creating the whole mouth score, the arithmatic average of all tooth scores was taken.
Attachment loss | Clinical periodontal indices were recorded at the participants' first visit.
  The scores from the four areas of the tooth are added and divided by four for each tooth score. It is recorded as mm. When creating the whole mouth score, the arithmatic average of all tooth scores was taken.
Bleeding on probing | Clinical periodontal indices were recorded at the participants' first visit.
  All four surfaces of all teeth are assessed with regard to whether probing elicits bleeding (+) or not (-).It is recorded as a percentage by umber of bleeding sites is number of sites evaluated and multiplying by one hundred.
Determination of GCF and Saliva SOST level | 1 month after all saliva and gingival crevicular fluid samples of the participants were collected between 01.12.2021-30.09.2022, SOST, TWEAK, RANKL and OPG levels were examined by ELISA method.
  Determination of SOST levels by ELISA method. It is recorded as pg/ml.
Determination of GCF and Saliva TWEAK level | 1 month after all saliva and gingival crevicular fluid samples of the participants were collected between 01.12.2021-30.09.2022, SOST, TWEAK, RANKL and OPG levels were examined by ELISA method.
  Determination of TWEAK levels by ELISA method. It is recorded as mg/l.
Determination of GCF RANKL level | 1 month after all saliva and gingival crevicular fluid samples of the participants were collected between 01.12.2021-30.09.2022, SOST, TWEAK, RANKL and OPG levels were examined by ELISA method.
  Determination of RANKL levels by ELISA method. It is recorded as pg/ml.
Determination of GCF OPG level | 1 month after all saliva and gingival crevicular fluid samples of the participants were collected between 01.12.2021-30.09.2022, SOST, TWEAK, RANKL and OPG levels were examined by ELISA method.
  Determination of OPG levels by ELISA method. It is recorded as pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Güner, Phd, Study Chair — Gazi University Faculty of Dentistry; Gülay Tüter, Professor, Study Director — Gazi University
Locations (1):
- Ece Güner, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gur AT, Guncu GN, Akman AC, Pinar A, Karabulut E, Nohutcu RM. Evaluation of GCF IL-17, IL-10, TWEAK, and sclerostin levels after scaling and root planing and adjunctive use of diode laser application in patients with periodontitis. J Periodontol. 2022 Aug;93(8):1161-1172. doi: 10.1002/JPER.21-0494. Epub 2022 Jan 25. PMID 34962665
- [Result] Rezaei Esfahrood Z, Yadegari Z, Veysari SK, Kadkhodazadeh M. Gingival crevicular fluid levels of sclerostin in chronic periodontitis and healthy subjects. J Korean Assoc Oral Maxillofac Surg. 2018 Dec;44(6):289-292. doi: 10.5125/jkaoms.2018.44.6.289. Epub 2018 Dec 28. PMID 30637243
- [Result] Teodorescu AC, Martu I, Teslaru S, Kappenberg-Nitescu DC, Goriuc A, Luchian I, Martu MA, Solomon SM, Martu S. Assessment of Salivary Levels of RANKL and OPG in Aggressive versus Chronic Periodontitis. J Immunol Res. 2019 Apr 28;2019:6195258. doi: 10.1155/2019/6195258. eCollection 2019. PMID 31183390

DOCUMENTS (3):
  • Study Protocol (2023-10-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT06103578/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT06103578/SAP_001.pdf
  • Informed Consent Form (2023-10-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT06103578/ICF_002.pdf